CLINICAL TRIAL: NCT01054573
Title: An Open-label, Single-arm, Roll-over Trial of Telaprevir in Combination With Pegylated Interferon Alfa-2a (Pegasys) and Ribavirin (Copegus) for Subjects From the Control Group of the VX- 950-TiDP24-C216 Trial Who Failed Therapy for Virologic Reasons
Brief Title: VX-950-TiDP24-C219: A Roll Over Trial for Patients in the Control Group of the C216 Study Who Received Telaprevir Placebo
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Infectious Diseases BVBA (Industry)
Collaborators: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR016678; VX-TiDP24-C219 (Other: Janssen Infectious Diseases BVBA); 2009-012613-21 (EudraCT Number)
Record Dates: First submitted 2010-01-21; First posted 2010-01-22 (Estimated); Results first posted 2013-04-19 (Estimated); Last update posted 2013-05-08 (Estimated); Status verified 2013-05

CONDITIONS: Hepatitis C, Chronic
Keywords: Hepatitis C, Chronic; Telaprevir; Roll-over study
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — telaprevir; peginterferon alfa-2a; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Telaprevir + Standard Treatment (Experimental): Telaprevir 750 mg orally (by mouth) every 8h for 12 weeks plus standard treatment. Standard treatment is 180 mcg subcutaneous (under the skin) injection pegylated interferon (Peg-IFN) alfa-2a and 1000-1200 mg twice daily ribavirin (RBV) for 48 weeks.
  Interventions: Drug: Telaprevir; Drug: pegylated interferon (Peg-IFN) alfa-2a; Drug: ribavirin (RBV)

INTERVENTIONS:
Drug: Telaprevir — 750 mg orally every 8 hours (q8h) for 12 weeks
Drug: pegylated interferon (Peg-IFN) alfa-2a — 180 microgram (mcg) by subcutaneous injection once weekly for 48 weeks.
Drug: ribavirin (RBV) — 1,000 or 1,200 mg/day (weight based) orally twice daily for 48 weeks.

SUMMARY:
The purpose of this study is to provide access to telaprevir for patients from the control group in the C216 study, who failed treatment for virologic reasons. Efficacy, safety and tolerability of telaprevir in combination with standard treatment will be evaluated.

DETAILED DESCRIPTION:
This is an open-label (i.e all people involved know the identity of the intervention), single-arm, roll-over trial of telaprevir in combination with pegylated interferon (Peg-IFN) alfa-2a and ribavirin (RBV). The purpose of the trial is to provide access to telaprevir for patients who were randomized to the control group in the VX-950-TiDP24-C216 trial (referred to as C216 trial hereafter) and who failed therapy for virologic reasons. The efficacy, safety, and tolerability of telaprevir in combination with Peg IFN alfa 2a and RBV will be evaluated. In addition, amino acid changes from baseline in the HCV NS3 (i.e protein associated with the hepatitis C virus) protease domain will be evaluated. The trial will consist of a screening period of approximately 28 days, a 48-week treatment period, and a 24-week follow-up period. It is expected that approximately 120 patients could be eligible for enrollment. Since the C216 trial is blinded until all patients reach Week 72 (or have discontinued earlier), patients can only enter the current trial upon invitation. The investigator will receive an invitation sent by the unblinded independent virology monitor of the C216 trial for those patients of the C216 trial who were randomized to the control group and who failed therapy for virologic reasons. Next to this invitation, the patient will need to fulfill the inclusion and exclusion criteria of the current trial in order to be eligible to participate. The screening visit for the current trial can only occur after the patient completes all assessments in the C216 trial, including the Safety Follow-up Visit. Patients must not enter this trial later than 80 weeks after their first dose in the C216 trial. In the current trial, all patients will receive 12 weeks of telaprevir 750 mg every 8 hours (q8h) in combination with Peg-IFN alfa-2a and RBV at standard doses, i.e., 180 microgram once weekly and 1,000 or 1,200 mg/day (weight based), respectively, followed by 36 weeks of Peg IFN alfa 2a and RBV at standard doses. Patients with hepatitis C virus RNA levels < 25 IU/mL undetectable at the end of treatment (Week 48 or having discontinued earlier) will be followed for 24 weeks after the last dose of study medication to assess sustained virologic response (SVR). Safety/tolerability assessments will be performed and adverse events (AEs), regardless of severity, will be collected continuously until the Safety Follow-up Visit, scheduled 4 weeks after the last dose of study medication. Thereafter, only serious adverse events (SAEs) will be reported. All patients will receive 12 weeks of telaprevir 750 mg q8h (orally) in combination with Peg-IFN alfa-2a and RBV at standard doses, i.e., 180 microgram once weekly (injection) and 1,000 or 1,200 mg/day (weight-based) (orally), respectively, followed by 36 weeks of Peg IFN alfa-2a and RBV at standard doses.

ELIGIBILITY:
Inclusion Criteria:

* Patient from the control group of the C216 study who failed therapy for virologic reasons
* Patient must have completed all assessments in the C216 trial
* Patient must be willing to use 2 effective methods of birth control for up to 7 months after last dose of study medication

Exclusion Criteria:

* Patient received any direct acting anti-viral HCV therapy after discontinuation of the C216 trial
* Patient has history of decompensated liver disease
* Patient has history of acute or chronic pancreatitis
* Patient has condition that requires use of systemic corticosteroids
* Patient who prematurely stopped medication for non-compliance or for whom it would be unsafe to repeat treatment
* Patient has history of decompensated liver disease or history of cirrhosis with hepatocellular carcinoma

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2010-04; Primary Completion 2012-03 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Infectious Diseases BVBA Clinical Trial, Study Director — Janssen Infectious Diseases BVBA
Locations (48):
- United States (14):
  - Coronado, California
  - Los Angeles, California
  - San Francisco, California
  - Bradenton, Florida
  - Miami, Florida
  - Atlanta, Georgia
  - Indianapolis, Indiana
  - Kansas City, Missouri
  - New York, New York
  - Chapel Hill, North Carolina
  - Philadelphia, Pennsylvania
  - Columbia, South Carolina
  - Houston, Texas
  - San Antonio, Texas
- Australia (4):
  - Adelaide
  - Clayton
  - Darlinghurst
  - Perth
- Belgium (3):
  - Brussels
  - Ghent
  - Leuven
- Brazil (3):
  - Distrito Barao Geraldo-Campina
  - Salvador
  - São Paulo
- Montreal, Quebec, Canada
- France (4):
  - Clichy
  - Créteil
  - Lille
  - Pessac
- Germany (6):
  - Berlin
  - Cologne
  - Frankfurt
  - Hamburg
  - Hanover
  - München
- Israel (2):
  - Petah Tikva
  - Safed
- Netherlands (2):
  - Amsterdam
  - Nijmegen
- Poland (3):
  - Bialystok
  - Czeladź
  - Warsaw
- San Juan, Puerto Rico
- Spain (2):
  - Barcelona
  - Valencia
- Stockholm, Sweden
- Zurich, Switzerland
- London, United Kingdom

REFERENCES:
- [Derived] Susser S, Flinders M, Reesink HW, Zeuzem S, Lawyer G, Ghys A, Van Eygen V, Witek J, De Meyer S, Sarrazin C. Evolution of hepatitis C virus quasispecies during repeated treatment with the NS3/4A protease inhibitor telaprevir. Antimicrob Agents Chemother. 2015 May;59(5):2746-55. doi: 10.1128/AAC.04911-14. Epub 2015 Feb 23. PMID 25712364

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 90 participants were enrolled and received treatment in the study: 9 participants from Phase 1 studies VX04-950-101 or Study VX05-950-103 and 81 participants from the Phase 3 study VX-950-TiDP24-C216 (NCT00703118) (referred to as the parent studies). The current study was conducted in 16 countries including the United States.
Pre-assignment Details: This study provided participants with access to telaprevir who were randomized to the control group in a previous Phase 3 study and failed therapy with pegylated interferon (Peg-IFN) alfa-2a and ribavirin (RBV) or to participants who received telaprevir as monotherapy or in combination with Peg-IFN-alfa-2a in 2 previous Phase 1 studies.
Groups:
- Phase 1: T12(Q8h)/PR: T12(Q8)/PR=Telaprevir every 8 hours for 12 weeks in combination with pegylated interferon (Peg-IFN) alfa-2a + ribavirin (RBV) administered for 48 weeks to participants who rolled-over from Phase 1 Studies VX04-950-101 or VX05-950-103.
- Phase 3: T12(Q8h)/PR - Prior Null Responder: T12(Q8)/PR=Telaprevir every 8 hours for 12 weeks in combination with pegylated interferon (Peg-IFN) alfa-2a + ribavirin (RBV) administered for 48 weeks to participants who rolled-over from Phase 3 Study VX-950-TiDP24-C216 (NCT00703118) control group who failed prior therapy due to virologic reasons and were categorized as prior null responders.
- Phase 3: T12(Q8h)/PR - Prior Partial Responder: T12(Q8)/PR=Telaprevir every 8 hours for 12 weeks in combination with pegylated interferon (Peg-IFN) alfa-2a + ribavirin (RBV) administered for 48 weeks to participants who rolled-over from Phase 3 Study VX-950-TiDP24-C216 (NCT00703118) control group who failed prior therapy for virologic reasons and were categorized as prior partial responders.
- Phase 3: T12(Q8h)/PR - Prior Relapser: T12(Q8)/PR=Telaprevir every 8 hours for 12 weeks in combination with pegylated interferon (Peg-IFN) alfa-2a + ribavirin (RBV) administered for 48 weeks to participants who rolled-over from Phase 3 Study VX-950-TiDP24-C216 (NCT00703118) control group who failed prior therapy for virologic reasons and were categorized as prior relapsers.
Period: Overall Study
Arm/Group | Phase 1: T12(Q8h)/PR | Phase 3: T12(Q8h)/PR - Prior Null Responder | Phase 3: T12(Q8h)/PR - Prior Partial Responder | Phase 3: T12(Q8h)/PR - Prior Relapser
Started | 9 | 32 | 22 | 27
Completed | 8 | 28 | 19 | 25
Not Completed | 1 | 4 | 3 | 2
Not completed — Adverse Event | 1 | 0 | 1 | 1
Not completed — Lost to Follow-up | 0 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 2 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1: T12(Q8h)/PR | Phase 3: T12(Q8h)/PR - Prior Null Responder | Phase 3: T12(Q8h)/PR - Prior Partial Responder | Phase 3: T12(Q8h)/PR - Prior Relapser | Total
Number analyzed (Participants) | 9 | 32 | 22 | 27 | 90
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 8 | 30 | 22 | 20 | 80
  >=65 years | 1 | 2 | 0 | 7 | 10
Age Continuous [Median (Inter-Quartile Range); unit: years] | 52 [49 to 61] | 51.5 [42 to 59.5] | 50.5 [47 to 58] | 55 [46 to 66] | 53 [45 to 60]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 9 | 7 | 8 | 28
  Male | 5 | 23 | 15 | 19 | 62
Region of Enrollment [Number; unit: participants]
  Europe | 9 | 18 | 10 | 14 | 51
  North America | 0 | 12 | 7 | 4 | 23
  Other | 0 | 2 | 5 | 9 | 16

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Participants Achieving a Sustained Virologic Response (SVR) 24 Weeks After the Last Dose of Study Drug (SVR24 Actual)
Description: The table below shows the percentage of participants acheiving a SVR 24 weeks after the last dose of study drug defined as having plasma hepatitis C virus (HCV) ribonucleic acid (RNA) levels < 25 IU/mL, target not detected at end of treatment (EOT) AND the participant did not relapse AND the participant completed the treatment; OR if the participant had plasma HCV RNA levels of < 25 IU/mL, target not detected at EOT AND the participant did not relapse AND the participant prematurely discontinued at least one study medication, but never for the reason virologic failure.
Time Frame: End of trial (24 weeks after last dose, administerd at 48 weeks)
Population: All analyses were performed on the full analysis (FA) set, which was defined as all randomized participants who received at least one dose of study drug.
Measure: Number; unit: Percentage of participants with response
Arm/Group | Phase 3: T12(Q8h)/PR - Prior Null Responder | Phase 3: T12(Q8h)/PR - Prior Partial Responder | Phase 3: T12(Q8h)/PR - Prior Relapser | Phase 1: T12(Q8h)/PR
Number analyzed (Participants) | 32 | 22 | 27 | 9
Percentage of participants with response | 34.4 | 72.7 | 81.5 | 44.4

2. Secondary Outcome: The Percentage of Participants Achieving Hepatitis C Virus (HCV) Ribonucleic Acid (RNA) Values of Less Than 25 IU/ml, Target Not Detected at Different Time Points
Description: The table below shows the percentage of participants with undetectable hepatitis C virus (HCV) ribonucleic acid (RNA) levels of less than 25 IU/ml, target not detected at different time points during the study. Data was imputed for participants with missing values using the last observation carried forward (LOCF) method for missing values.
Time Frame: Baseline, Weeks 4, 8, 12, 24, 36, and 48, and at the end of treatment (Week 48 or at time of early discontinuation)
Population: as for outcome 1
Measure: Number; unit: Percentage of participants with response
Arm/Group | Phase 3: T12(Q8h)/PR - Prior Null Responder | Phase 3: T12(Q8h)/PR - Prior Partial Responder | Phase 3: T12(Q8h)/PR - Prior Relapser | Phase 1: T12(Q8h)/PR
Number analyzed (Participants) | 32 | 22 | 27 | 9
Percentage of participants with response
  Basline | 0 | 0 | 0 | 0
  Week 4 | 37.5 | 77.3 | 85.2 | 33.3
  Week 8 | 56.3 | 86.4 | 92.6 | 66.7
  Week 12 | 59.4 | 90.9 | 92.6 | 66.7
  Week 24 | 50.0 | 77.3 | 85.2 | 66.7
  Week 36 | 43.8 | 81.8 | 85.2 | 77.8
  Week 48 | 43.8 | 72.7 | 85.2 | 77.8
  End of Treatment | 43.8 | 86.4 | 92.6 | 77.8

3. Secondary Outcome: Percentage of Participants Who Met a Virologic Stopping Rule That Required Them to Permanently Discontinue Telaprevir and Continue Pegylated Interferon (Peg-IFN) and Ribavirin (RBV) at Week 4 or Week 8
Description: The table below shows the percentage of participants at Week 4 or 8 who met a stopping rule defined as having a hepatitis C virus (HCV) ribonucleic acid (RNA) value >100 IU/mL.
Time Frame: Week 4, Week 8
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Groups:
- Phase 3: T12(Q8h)/PR - Prior Null Responder: T12(Q8)/PR=Telaprevir every 8 hours for 12 weeks in combination with pegylated interferon (Peg-IFN) alfa-2a + ribavirin (RBV) administered for 48 weeks to participants who rolled-over from Phase 3 Study VX-950-TiDP24-C216(NCT00703118) control group who failed prior therapy due to virologic reasons and were categorized as prior null responders.
Arm/Group | Phase 3: T12(Q8h)/PR - Prior Null Responder | Phase 3: T12(Q8h)/PR - Prior Partial Responder | Phase 3: T12(Q8h)/PR - Prior Relapser | Phase 1: T12(Q8h)/PR
Number analyzed (Participants) | 32 | 22 | 27 | 9
Percentage of participants | 28.1 | 4.5 | 3.7 | 11.1

4. Secondary Outcome: Percentage of Participants Who Met a Virologic Stopping Rule That Required Them to Permanently Discontinue All Study Drugs at Week 12, 24, or 36
Description: The table below shows the percentage of participants at Week 12, 24, and 36 who met a stopping rule. The stopping rule at Week 12 was having hepatitis C virus (HCV) ribonucleic acid (RNA) value of >100 IU/mL and the stopping rule at Weeks 24 or 36 was having a HCV RNA value of >=25 IU/mL.
Time Frame: Week 12 or Weeks 24 or 36
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Groups:
- Phase 3: T12(Q8h)/PR - Prior Partial Responder: T12(Q8)/PR=Telaprevir every 8 hours for 12 weeks in combination with pegylated interferon (Peg-IFN) alfa-2a + ribavirin (RBV) administered for 48 weeks to participants who rolled-over from Phase 3 Study VX-950-TiDP24-C216(NCT00703118) control group who failed prior therapy for virologic reasons and were categorized as prior partial responders.
- Phase 3: T12(Q8h)/PR - Prior Relapser: T12(Q8)/PR=Telaprevir every 8 hours for 12 weeks in combination with pegylated interferon (Peg-IFN) alfa-2a + ribavirin (RBV) administered for 48 weeks to participants who rolled-over from Phase 3 Study VX-950-TiDP24-C216(NCT00703118) control group who failed prior therapy for virologic reasons and were categorized as prior relapsers.
Arm/Group | Phase 3: T12(Q8h)/PR - Prior Null Responder | Phase 3: T12(Q8h)/PR - Prior Partial Responder | Phase 3: T12(Q8h)/PR - Prior Relapser | Phase 1: T12(Q8h)/PR
Number analyzed (Participants) | 32 | 22 | 27 | 9
Percentage of participants
  Week 12 | 31.2 | 4.5 | 0 | 11.1
  Week 24 | 9.4 | 9.1 | 3.7 | 11.1
  Week 36 | 9.4 | 0 | 0 | 0

5. Secondary Outcome: Percentage of Participants Achieving Rapid Virologic Response (RVR)
Description: The table below shows the percentage of participants who had a rapid virologic response (RVR) (ie, those with undetectable hepatitis C virus [HCV] ribonucleic acid [RNA values of <25 IU/mL, target not detected at Week 4 of treatment).
Time Frame: Week 4
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Phase 3: T12(Q8h)/PR - Prior Null Responder | Phase 3: T12(Q8h)/PR - Prior Partial Responder | Phase 3: T12(Q8h)/PR - Prior Relapser | Phase 1: T12(Q8h)/PR
Number analyzed (Participants) | 32 | 22 | 27 | 9
Percentage of participants | 37.5 | 77.3 | 85.2 | 33.3

6. Secondary Outcome: Percentage of Participants Achieving Extended Rapid Virologic Response (eRVR)
Description: The table below shows the percentage of participants who had a Extended Rapid Virologic Response (eRVR) (ie, those with undetectable hepatitis C virus [HCV] ribonucleic acid [RNA values of <25 IU/mL, target not detected at at Weeks 4 and 12 of treatment).
Time Frame: Weeks 4 and 12
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Phase 3: T12(Q8h)/PR - Prior Null Responder | Phase 3: T12(Q8h)/PR - Prior Partial Responder | Phase 3: T12(Q8h)/PR - Prior Relapser | Phase 1: T12(Q8h)/PR
Number analyzed (Participants) | 32 | 22 | 27 | 9
Percentage of participants | 34.4 | 72.7 | 85.2 | 33.3

7. Secondary Outcome: Percentage of Participants With Viral Breakthrough
Description: The table below shows the percentage of participants with viral breakthrough defined as a confirmed increase >1 log10 in hepatitis C virus (HCV) ribonucleic acid (RNA) level from the lowest level reached during the considered treatment phase up to the considered time point, if the lowest level reached is > 25 IU/mL, or a confirmed value of HCV RNA >100 IU/mL in participants whose HCV RNA had previously become <25 IU/mL (detected or target not detected) during the considered treatment phase.
Time Frame: Week 48 (Period After Telaprevir Intake) and Week 12 (Telaprevir Treatment Phase)
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Phase 3: T12(Q8h)/PR - Prior Null Responder | Phase 3: T12(Q8h)/PR - Prior Partial Responder | Phase 3: T12(Q8h)/PR - Prior Relapser | Phase 1: T12(Q8h)/PR
Number analyzed (Participants) | 32 | 22 | 27 | 9
Percentage of participants
  Week 48 (Period After Telaprevir Intake) | 25.0 | 9.1 | 3.7 | 11.1
  Week 12 (Telaprevir Treatment Phase) | 15.6 | 4.5 | 0.0 | 11.1

8. Secondary Outcome: Percentage of Participants Who Relapsed During Follow-Up
Description: The table below shows the percentage of participants who relapsed (ie, those having confirmed detectable hepatitis C virus [HCV] ribonucleic acid [RNA] during the 24-week follow-up period after previous HCV RNA <25 IU/mL, target not detected, at end of treatment).
Time Frame: During Follow-Up (24 weeks after the last dose of study drug, administerd at 48 weeks)
Population: The analysis was performed on the full analysis (FA) set, which included all randomized participants who received at least one dose of study drug and had data at the follow-up visit performed 24 weeks after the last dose of study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Phase 3: T12(Q8h)/PR - Prior Null Responder | Phase 3: T12(Q8h)/PR - Prior Partial Responder | Phase 3: T12(Q8h)/PR - Prior Relapser | Phase 1: T12(Q8h)/PR
Number analyzed (Participants) | 14 | 19 | 25 | 7
Percentage of participants | 21.4 | 5.3 | 4.0 | 28.6

9. Secondary Outcome: Hepatitis C Virus (HCV) Ribonucleic Acid (RNA) Values Over Time
Description: The table below shows plasma Hepatitis C virus (HCV) ribonucleic acid (RNA) values measured over time.
Time Frame: Baseline, Weeks 4, 8, 12, 24, 36, 48
Population: as for outcome 1
Measure: Median (Full Range); unit: Log 10 IU/mL
Groups:
- Phase 3: T12(Q8h)/PR - Prior Null Responder: T12(Q8)/PR=Telaprevir every 8 hours for 12 weeks in combination with pegylated interferon (Peg-IFN) alfa-2a + ribavirin (RBV) administered for 48 weeks to participants who rolled-over from Phase 3 Study VX-950-TiDP24-C216(NCT00703118) control group who failed prior therapy due to virologic reasons and were categorized as prior null responders. The number of participants analyzed at Baseline and Weeks 4, 8, 12, 24, 36, and 48 were: 32, 32, 32, 31, 23, 18, and 16, respectively.
- Phase 3: T12(Q8h)/PR - Prior Partial Responder: T12(Q8)/PR=Telaprevir every 8 hours for 12 weeks in combination with pegylated interferon (Peg-IFN) alfa-2a + ribavirin (RBV) administered for 48 weeks to participants who rolled-over from Phase 3 Study VX-950-TiDP24-C216(NCT00703118) control group who failed prior therapy for virologic reasons and were categorized as prior partial responders. The number of participants analyzed at Baseline and Weeks 4, 8, 12, 24, 36, and 48 were: 22, 22, 22, 22, 20, 19, and 16, respectively.
- Phase 3: T12(Q8h)/PR - Prior Relapser: T12(Q8)/PR=Telaprevir every 8 hours for 12 weeks in combination with pegylated interferon (Peg-IFN) alfa-2a + ribavirin (RBV) administered for 48 weeks to participants who rolled-over from Phase 3 Study VX-950-TiDP24-C216(NCT00703118) control group who failed prior therapy for virologic reasons and were categorized as prior relapsers. The number of participants analyzed at Baseline and Weeks 4, 8, 12, 24, 36, and 48 were: 27, 26, 26, 26, 24, 23, and 21, respectively.
- Phase 1: T12(Q8h)/PR: T12(Q8)/PR=Telaprevir every 8 hours for 12 weeks in combination with pegylated interferon (Peg-IFN) alfa-2a + ribavirin (RBV) administered for 48 weeks to participants who rolled-over from Phase 1 Studies VX04-950-101 or VX05-950-103. The number of participants analyzed at Baseline and Weeks 4, 8, 12, 24, 36, and 48 were: 9, 9, 9, 9, 9, 8, 7, and 7, respectively.
Arm/Group | Phase 3: T12(Q8h)/PR - Prior Null Responder | Phase 3: T12(Q8h)/PR - Prior Partial Responder | Phase 3: T12(Q8h)/PR - Prior Relapser | Phase 1: T12(Q8h)/PR
Number analyzed (Participants) | 32 | 22 | 27 | 9
Log 10 IU/mL
  Baseline (n=32, 22, 27, and 9) | 6.63 [5.2 to 7.3] | 6.72 [5.6 to 7.3] | 6.48 [5.3 to 7.5] | 6.76 [6.0 to 7.2]
  Week 4 (n=32, 22, 26, and 9) | 1.24 [0.7 to 6.7] | 0.70 [0.7 to 1.2] | 0.70 [0.7 to 2.3] | 1.24 [0.7 to 1.5]
  Week 8 (n=32, 22, 26, and 9) | 0.70 [0.7 to 6.9] | 0.70 [0.7 to 2.7] | 0.70 [0.7 to 1.6] | 0.70 [0.7 to 2.9]
  Week 12 (n=31, 22, 26, and 9) | 0.70 [0.7 to 7.1] | 0.70 [0.7 to 4.3] | 0.70 [0.7 to 1.2] | 0.70 [0.7 to 5.5]
  Week 24 (n=23, 20, 26, and 8) | 0.70 [0.7 to 6.6] | 0.70 [0.7 to 4.8] | 0.70 [0.7 to 2.1] | 0.70 [0.7 to 6.2]
  Week 36 (n=18, 19, 23, and 7) | 0.70 [0.7 to 4.8] | 0.70 [0.7 to 4.8] | 0.70 [0.7 to 0.7] | 0.70 [0.7 to 0.7]
  Week 48 (n=16, 16, 21, and 7) | 0.70 [0.7 to 2.3] | 0.70 [0.7 to 0.7] | 0.70 [0.7 to 0.7] | 0.70 [0.7 to 0.7]

10. Secondary Outcome: Change From Baseline in Log 10 Plasma Hepatitis C Virus (HCV) Ribonucleic Acid (RNA) Level
Description: The table below shows change from baseline in log 10 plasma HCV RNA values measured over time.
Time Frame: Baseline, Weeks 4, 8, 12, 24, 36, and 48
Population: as for outcome 1
Measure: Median (Full Range); unit: log 10 IU/ml
Groups:
- Phase 3: T12(Q8h)/PR - Prior Null Responder: T12(Q8)/PR=Telaprevir every 8 hours for 12 weeks in combination with pegylated interferon (Peg-IFN) alfa-2a + ribavirin (RBV) administered for 48 weeks to participants who rolled-over from Phase 3 Study VX-950-TiDP24-C216(NCT00703118) control group who failed prior therapy due to virologic reasons and were categorized as prior null responders. The number of participants analyzed at Weeks 4, 8, 12, 24, 36, and 48 were: 32, 32, 31, 23, 18, and 15, respectively.
- Phase 3: T12(Q8h)/PR - Prior Partial Responder: T12(Q8)/PR=Telaprevir every 8 hours for 12 weeks in combination with pegylated interferon (Peg-IFN) alfa-2a + ribavirin (RBV) administered for 48 weeks to participants who rolled-over from Phase 3 Study VX-950-TiDP24-C216(NCT00703118) control group who failed prior therapy for virologic reasons and were categorized as prior partial responders. The number of participants analyzed at Weeks 4, 8, 12, 24, 36, and 48 were: 22, 22, 22, 20, 19, and 16, respectively.
- Phase 3: T12(Q8h)/PR - Prior Relapser: T12(Q8)/PR=Telaprevir every 8 hours for 12 weeks in combination with pegylated interferon (Peg-IFN) alfa-2a + ribavirin (RBV) administered for 48 weeks to participants who rolled-over from Phase 3 Study VX-950-TiDP24-C216(NCT00703118) control group who failed prior therapy for virologic reasons and were categorized as prior relapsers. The number of participants analyzed at Weeks 4, 8, 12, 24, 36, and 48 were: 26, 26, 26, 24, 23, and 21, respectively.
- Phase 1: T12(Q8h)/PR: T12(Q8)/PR=Telaprevir every 8 hours for 12 weeks in combination with pegylated interferon (Peg-IFN) alfa-2a + ribavirin (RBV) administered for 48 weeks to participants who rolled-over from Phase 1 Studies VX04-950-101 or VX05-950-103. The number of participants analyzed at Weeks 4, 8, 12, 24, 36, and 48 were: 9, 9, 9, 8, 7, and 7, respectively.
Arm/Group | Phase 3: T12(Q8h)/PR - Prior Null Responder | Phase 3: T12(Q8h)/PR - Prior Partial Responder | Phase 3: T12(Q8h)/PR - Prior Relapser | Phase 1: T12(Q8h)/PR
Number analyzed (Participants) | 32 | 22 | 27 | 9
log 10 IU/ml
  Week 4 (n=32, 22, 26, and 9) | -5.39 [-6.6 to -0.6] | -5.83 [-6.6 to -4.9] | -5.59 [-6.8 to -4.4] | -5.55 [-6.1 to -5.1]
  Week 8 (n=32, 22, 26, and 9) | -5.51 [-6.6 to -0.4] | -5.88 [-6.6 to -4.6] | -5.62 [-6.8 to -4.6] | -5.96 [-6.3 to -3.4]
  Week 12 (n=31, 22, 26, 9) | -5.40 [-6.6 to -0.2] | -5.88 [-6.6 to -3.0] | -5.62 [-6.8 to -4.6] | -5.96 [-6.3 to -0.9]
  Week 24 (n=23, 20, 24, and 8) | -5.89 [-6.6 to 1.0] | -5.72 [-6.6 to -2.2] | -5.75 [-6.8 to -4.6] | -5.87 [-6.1 to -1.0]
  Week 36 (n=18, 19, 23, and 7) | -5.95 [-6.6 to -0.6] | -5.86 [-6.6 to -2.3] | -5.78 [-6.8 to -4.6] | -6.07 [-6.3 to -5.3]
  Week 48 (n=15, 16, 21, and 7) | -6.03 [-6.6 to -4.1] | -5.88 [-6.6 to -5.2] | -5.71 [-6.8 to -4.6] | -6.07 [-6.3 to -5.3]

ADVERSE EVENTS:
Time Frame: From Baseline (Day 1) through Week 48 (or last dose of study drug received) + 24 week follow-up period.
Groups:
- Phase 3: T12(Q8h)/PR: T12(Q8)/PR=Telaprevir every 8 hours for 12 weeks in combination with pegylated interferon (Peg-IFN) alfa-2a + ribavirin (RBV) administered for 48 weeks to participants who rolled-over from Phase 3 Study VX-950-TiDP24-C216(NCT00703118) control group who failed prior therapy due to virologic reasons (ncludes all participants, ie, those categorized as prior null responders, prior partial responders, and prior relapsers).
Arm/Group | Phase 1: T12(Q8h)/PR | Phase 3: T12(Q8h)/PR
Serious Adverse Events (participants affected / at risk) | 0/9 | 5/81
Other Adverse Events (participants affected / at risk) | 9/9 | 77/81
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1: T12(Q8h)/PR (N=9) | Phase 3: T12(Q8h)/PR (N=81)
Anaemia (Blood and lymphatic system disorders) | 0 | 3
Biliary colic (Hepatobiliary disorders) | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1: T12(Q8h)/PR (N=9) | Phase 3: T12(Q8h)/PR (N=81)
Anaemia (Blood and lymphatic system disorders) | 1 | 23
Leukopenia (Blood and lymphatic system disorders) | 0 | 8
Neutropenia (Blood and lymphatic system disorders) | 1 | 11
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 7
Vertigo (Ear and labyrinth disorders) | 1 | 1
Dry eye (Eye disorders) | 1 | 1
Anal pruritus (Gastrointestinal disorders) | 0 | 6
Anorectal discomfort (Gastrointestinal disorders) | 0 | 6
Aphthous stomatitis (Gastrointestinal disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 12
Dry mouth (Gastrointestinal disorders) | 0 | 5
Dyspepsia (Gastrointestinal disorders) | 0 | 5
Gastritis (Gastrointestinal disorders) | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 9
Nausea (Gastrointestinal disorders) | 5 | 18
Vomiting (Gastrointestinal disorders) | 1 | 5
Asthenia (General disorders) | 0 | 15
Fatigue (General disorders) | 7 | 33
Influenza like illness (General disorders) | 3 | 8
Irritability (General disorders) | 0 | 10
Mucosal inflammation (General disorders) | 1 | 0
Pyrexia (General disorders) | 0 | 11
Bronchitis (Infections and infestations) | 1 | 0
Cystitis (Infections and infestations) | 1 | 1
Fungal infection (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 2
Upper respiratory tract infection (Infections and infestations) | 1 | 2
Weight decreased (Investigations) | 0 | 5
Anorexia (Metabolism and nutrition disorders) | 0 | 5
Decreased appetite (Metabolism and nutrition disorders) | 0 | 12
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 7
Disturbance in attention (Nervous system disorders) | 1 | 2
Dizziness (Nervous system disorders) | 1 | 9
Headache (Nervous system disorders) | 3 | 17
Depression (Psychiatric disorders) | 3 | 6
Insomnia (Psychiatric disorders) | 1 | 12
Genital rash (Reproductive system and breast disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 9
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 9
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 5
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 2 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 9
Prurigo (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 33
Rash (Skin and subcutaneous tissue disorders) | 3 | 17
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 | 1
Hypertension (Vascular disorders) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
It is the policy of the sponsor not to allow the investigators to publish their results or findings prior to the sponsor's publication of the overall trial results. The investigator agrees that before he/she publishes any results of this trial, he/she shall allow at least 45 days for the sponsor to review the prepublication manuscript prior to submission of the manuscript to the publisher as specified in the Clinical Trial Agreement between institution/investigator and sponsor.